CLINICAL TRIAL: NCT00900822
Title: Randomized, Controlled Clinical Study to Compare Bone Formation Around Micro-implants in the Maxilla After Sinus Floor Augmentation With Straumann Bone Ceramic or Bio-Oss in a Split Mouth Design
Brief Title: Straumann Bone Ceramic Versus BioOss in Sinus Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 02/05
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Jaw, Edentulous, Partially; Alveolar Bone Loss
Keywords: bone grafting; sinus elevation; sinus augmentation
MeSH Terms: conditions — Jaw, Edentulous, Partially; Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Straumann Bone Ceramic (Experimental): StraumannBone Ceramic is used as bone grafting material in sinus augmentation procedures
  Interventions: Device: Straumann Bone Ceramic
- BioOss (Active Comparator): BioOss is used as a bone grafting material in sinus augmentation procedure
  Interventions: Device: BioOss

INTERVENTIONS:
Device: Straumann Bone Ceramic — Granules applied once during surgery
  Arms: Straumann Bone Ceramic
Device: BioOss — Granules that are applied once during surgery
  Arms: BioOss

SUMMARY:
Straumann Bone Ceramic (SBC) and BioOss will be used as bone grafting materials when there is a need for bone augmentation in the posterior upper jaw. 9 months later the bone formation is evaluated. The patients are followed for 3 years.The study hypothesis is that the SBC is not worse than BioOss.

DETAILED DESCRIPTION:
Straumann Bone Ceramic (SBC) and BioOss will be used as bone grafting materials when there is a need for bone augmentation in the posterior upper jaw. The bone grafting materials will be placed into the sinus cavity,(a routine procedure), one material randomly at each side and a micro-implant will be inserted simultaneously. 9 months later the micro-implant is removed and a regular Straumann SLActive implant is inserted. The micro-implant is evaluated histologically. The site is evaluated every 12 months for 3 years in regards to clinical measurements. The study hypothesis is that the SBC is not worse than BioOss.

Study design: Prospective, randomized, open, controlled, single center, split mouth

Study population: 11 male and female patients at an age of between 18 and 80 years, affected by edentulism of both lateral-posterior maxilla and presenting two pneumatized maxillary sinuses and necessitating rehabilitation with implant-supported prostheses will be recruited in the study and treated by means of maxillary sinus floor augmentation and delayed implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years to 80 years of age
* The patients are at least partly edentulous in the both maxillary regions corresponding to the sinuses.
* A dental implant procedure is foreseen in both maxilla regions corresponding to maxillary sinuses.
* Patients must be expected to present a bilateral bone defect in the sinus area, which both need a sinus floor augmentation to place one or more dental implants each.
* Residual alveolar crest height of the lateral-posterior segments of the edentulous maxilla below the floor of each of the maxillary sinuses shall be
* less than 5 mm and at least 2 mm, as measured by Scanora - tomography Scans in the deepest floor of the sinus
* residual alveolar crest width should be at least in average more than 4mm as measured by Scanora - tomography scans
* Patients must be committed to the study and must sign informed consent.
* Oral hygiene Index less than 25%

Exclusion Criteria:

* Any systemic medical condition that could interfere with the surgical procedure or planned treatment
* Current pregnancy at the time of recruitment
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Alcoholism or chronically drug abuse causing systemic compromize
* Patients who smoke more than 10 cigarettes per day
* Medication which interferes with bone formation
* Conditions or circumstances, in the opinion of the investigator, which could represent a general contra-indication for surgical procedure or would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability
* Mucosal diseases such as erosive lichen planus
* History of local radiation therapy
* Presence of oral lesions (such as ulceration, malignancy)
* Severe bruxing or clenching habits
* Persistent intraoral infection
* Previous GBR (bone graft) or dental implant treatment in the posterior segments of the upper maxilla (foreseen implant site)
* Patients presenting clinical and radiological signs and symptoms of maxillary sinus disease
* Existing teeth in the residual dentition with untreated endodontic problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mats Hallman, DDS, PhD, Principal Investigator — Clinic for oral maxillofacial surgery, Gävle hospital, Sweden
Locations (1):
- Dr Mats Hallman, Gävle, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lindgren C, Mordenfeld A, Hallman M. A prospective 1-year clinical and radiographic study of implants placed after maxillary sinus floor augmentation with synthetic biphasic calcium phosphate or deproteinized bovine bone. Clin Implant Dent Relat Res. 2012 Mar;14(1):41-50. doi: 10.1111/j.1708-8208.2010.00224.x. Epub 2010 May 11. PMID 20491816
- [Result] Lindgren C, Sennerby L, Mordenfeld A, Hallman M. Clinical histology of microimplants placed in two different biomaterials. Int J Oral Maxillofac Implants. 2009 Nov-Dec;24(6):1093-100. PMID 20162114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started Oct 2005 and was completed June 2006.
Pre-assignment Details: Split-mouth design (test and control in the same patient).
Groups:
- Straumann BoneCeramic: Synthetic bone graft material
Period: 9 Months Histological Evaluation
Arm/Group | Straumann BoneCeramic
Started | 11
Completed | 11
Not Completed | 0
Period: 12 Months Clinical Evaluation
Arm/Group | Straumann BoneCeramic
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Straumann Bone Ceramic: Synthetic bone graft material
Arm/Group | Straumann Bone Ceramic
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.27 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  Sweden | 11

OUTCOME MEASURES:

1. Secondary Outcome: Implant Survival Rate
Description: The percentage of implants remaining in the jaw.
Time Frame: 12 months after loading the implant
Measure: Number; unit: percentage of implants
Groups:
- BioOss: Xenograft bone graft material
Arm/Group | Straumann Bone Ceramic | BioOss
Number analyzed (Participants) | 11 | 11
percentage of implants | 96.7 | 96.7

2. Primary Outcome: Histologically Measured Bone to Implant Contact (BIC)
Description: Results from morphometric measurements of percentage of new bone in contact with the total surface of the titanium implant, area of new bone and bone graft particles in contact with bone
Time Frame: 9 months after implant placement
Population: This was a split-mouth design. Each patient received both treatments. There was one sample in the Straumann BoneCeramic group that could not be analyzed.
Measure: Mean (Standard Deviation); unit: percentage of total surface
Arm/Group | Straumann BoneCeramic | BioOss
Number analyzed (Participants) | 10 | 11
percentage of total surface | 64.552 (9.036) | 54.904 (15.995)

3. Secondary Outcome: Implant Success Rate
Description: Implant success is defined as the absence of any continuous peri-implant radiolucency based on radiographic findings, absence of implant mobility, absence of a recurrent per-implant infection with suppuration (where an infection is termed recurrent if it is observed at two or more 3-month follow-up visits after treatment with systemic antibiotics), and bone level changes around the implant less than 1 mm during the first year of loading and less than 0.2 mm per year thereafter.
Time Frame: 12 months after loading the implant
Measure: Number; unit: percentage of implants
Arm/Group | Straumann Bone Ceramic | BioOss
Number analyzed (Participants) | 11 | 11
percentage of implants | 93.6 | 96.8

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Straumann Bone Ceramic | BioOss
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 3/11 | 4/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Straumann Bone Ceramic (N=11) | BioOss (N=11)
Exposure of implant (General disorders) | 1 (1) | 1 (1)
Implant infection (General disorders) | 1 (1) | 0 (0)
Mobile implant (General disorders) | 0 (0) | 1 (1)
Fenestration of implant (General disorders) | 0 (0) | 1 (1)
Sinusitis (General disorders) | 1 (1) | 0 (0)
Contact between cover screw and prosthesis (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No